CLINICAL TRIAL: NCT04695522
Title: Phase I Trial of ADR-002K for Patients With Ischemic Cardiomyopathy Who Undergo Coronary Artery Bypass Surgery
Brief Title: ADR-002K for Patients With Ischemic Cardiomyopathy Who Undergo Coronary Artery Bypass Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osaka University (Other)
Collaborators: Rohto Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Daisuke Mori, Assistant professor, Osaka University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVSR0006
Record Dates: First submitted 2020-12-09; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: D017202
Keywords: Coronary artery bypass; Ischemic cardiomyopathy; Adipose-derived mesenchymal stem cells; Regenerative medicine; Spray method

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of subjects undergoing cell transplantation (Experimental)
  Interventions: Biological: ADR-002K administration
- Group of subjects undergoing sham operation (Sham Comparator)
  Interventions: Biological: ADR-002K administration

INTERVENTIONS:
Biological: ADR-002K administration — ADR-002K administration

SUMMARY:
Ischemic cardiomyopathy undergoing coronary artery bypass surgery

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are clinically diagnosed with ischemic cardiomyopathy and receive CABG
2. Patients with a left ventricular ejection fraction of 40% or less by cardiac ultrasonography within 4 weeks before obtaining consent
3. Others

Exclusion Criteria:

1. Patients who have a combination of cardiovascular disease such as severe organic valvular disease or aortic aneurysm determined by investigator or co-investigator to affect clinical trial procedure
2. Patients whose participation in a clinical trial is considered inappropriate at the discretion of the investigator or co-investigator
3. Others

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse event | 26 weeks
  Safety assessment related to adverse events and this product
Amount of change in late gadolinium contrast-enhanced area at the time of screening and 6 months after surgery | 26 weeks
  Efficacy (Exploratory)
Number of complication associated with drug administration method | 26 weeks
  Feasibility of drug administration method

CONTACTS AND LOCATIONS:
Overall Officials: Daisuke Mori, Ph.D, Principal Investigator — Osaka University Hospital
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kawamura T, Yoshioka D, Kawamura A, Misumi Y, Taguchi T, Mori D, Saito S, Yamauchi T, Hata H, Miyagawa S. Safety and therapeutic potential of allogeneic adipose-derived stem cell spray transplantation in ischemic cardiomyopathy: a phase I clinical trial. J Transl Med. 2024 Dec 2;22(1):1091. doi: 10.1186/s12967-024-05816-1. PMID 39623426